CLINICAL TRIAL: NCT02949700
Title: A Phase I/II Study OF Metformin in Combination With Cisplatin and Radiation in Head and Neck Squamous Cell Carcinoma
Brief Title: Phase I/II Study OF Metformin in Combination With Cisplatin and Radiation in Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Vlad Sandulache, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-39773
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Results first posted 2022-07-21 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: metformin; head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm, treatment (Experimental): Patients in the Phase I trial will be assigned to a single arm, experimental treatment which will test dose escalation for metformin in the context of chemo-radiation, with toxicity as the primary outcome.
  Patients in the Phase II trial will be assigned to a single arm, experimental treatment consisting of metformin plus chemo-radiation.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin will be administered orally twice daily during treatment with chemo-radiation for head and neck squamous cell carcinoma. This will occur 7 to 11 days prior to chemotherapy and radiation.

SUMMARY:
The purpose of this research is to see whether metformin can improve the response rate in patients undergoing chemotherapy and radiation for squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx. The purpose of this research is also to see the effects, good and bad, of metformin therapy for this disease. Researchers will also analyze tumor and blood samples from study patients to test and understand the characteristics of tumors which respond to metformin.

DETAILED DESCRIPTION:
Information from laboratory studies and retrospective studies of patients with this disease has shown that the addition of metformin (a commonly used medicine for treating diabetes) to chemotherapy and radiation can improve the rate at which the cancer responds to treatment. Metformin is used frequently in the treatment of patients with diabetes and other illness, but has not yet been used to treat patients with this type of cancer. In this research study, we want to see if using metformin during treatment with chemotherapy and radiation will increase the chance that the cancer will respond to treatment and not return.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Diagnosis: Patients must have histologically or cytologically confirmed squamous cell carcinoma (SCC) of the oral cavity, oropharynx, hypopharynx or larynx. Patients eligible for inclusion must have stage III-IV SCC of the above sites based on current AJCC clinical and imaging based staging (see Appendix A for staging criteria). For the phase II component, patients should present with: 1) HPV- SCC or 2) HPV+ SCC and a concomitant ≥10pack-year smoking history documented in the clinical record; HPV status will be ascertained using the currently utilized clinical standard of p16 overexpression via immunohistochemistry for all patients. Immunohistochemistry to determine p16 overexpression is only a requirement for oropharyngeal disease.
2. Disease Status: Only patients with active, measurable disease will be included in the study.
3. Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. Patients treated with chemotherapy (i.e. cisplatin) and/or EBRT for a cancer at a different, non-head and neck site, will be eligible for the trial. Patients previously treated with chemotherapy and/or EBRT for a cancer of the head and neck region, irrespective of histology will not be eligible to participate in the trial.
4. Myelosuppressive chemotherapy: Must not have received within 4 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
5. Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor.
6. Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent.
7. Monoclonal Antibody: At least 6 weeks must have elapsed since prior therapy that includes a monoclonal antibody.

   Other: For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
8. XRT: >/= 14days for local palliative XRT (small port); >/= 90days must have elapsed if prior TBI, craniospinal XRT or if >/= 50% radiation of pelvis; >/= 45days must have elapsed if other substantial bone marrow radiation.
9. Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and >/= 2 months must have elapsed since transplant.
10. Age: Patients must be >/=18 years of age. Because no dosing or adverse event data are currently available on the use of metformin in cancer patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
11. Performance Status: ECOG performance status less than or equal to 3.
12. Organ Function: Patients must have normal organ and marrow function as defined below:

    1. leukocytes >/= 3,000/mcL
    2. absolute neutrophil count >/= 1,500/mcL
    3. platelets >/= 100,000/mcL
    4. total bilirubin within normal institutional limits
    5. AST(SGOT) </= 2.5X institutional upper limit of normal
    6. creatinine < 1.5mg/dL OR
    7. creatinine clearance >/= 60 mL/min/1.73 m2 for patients with creatinine levels > institutional normal
13. Patients must be candidates for standard of care treatment consisting of chemotherapy (cisplatin) and radiation.
14. Willingness to Use Contraception: The effects of metformin on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
15. Informed Consent: Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Concomitant Medications: Patients may not be receiving any other investigational agents.
2. Brain metastases: Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
3. Prior Allergies: History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin.
4. Patients with diabetes mellitus (DM) will be excluded from the study. Criteria for a diagnosis of diabetes mellitus are as follows: a) known diagnosis of DM, b) active treatment for DM, c) fasting glucose level ≥ 126mg/dl or d) hemoglobin A1c ≥ 6.0% obtained within 30 days prior to registration.
5. Intercurrent Illness: Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Pregnancy: Patients may not be pregnant or breastfeeding.
7. HIV: HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with metformin. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
8. Patients taking metformin for any reason will not be eligible for inclusion in the study.
9. Patients may not have been treated for another SCC of the oral cavity, oropharynx, hypopharynx or larynx in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Sandulache, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kemnade JO, Florez M, Sabichi A, Zhang J, Jhaveri P, Chen G, Chen A, Miller-Chism C, Shaun B, Hilsenbeck SG, Hernandez DJ, Skinner HD, Sandulache VC. Phase I / II trial of metformin as a chemo-radiosensitizer in a head and neck cancer patient population. Oral Oncol. 2023 Oct;145:106536. doi: 10.1016/j.oraloncology.2023.106536. Epub 2023 Aug 8. PMID 37562095

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject withdrew consent prior to being assigned to a dose level. Therefore, 25 patients were assigned dose levels and began treatment.
Groups:
- Single Arm, Treatment: DL1 (Phase I); Single Arm, Treatment: DL1 (Phase II): Patients in the Phase I trial will be assigned to a single arm, experimental treatment which will test dose escalation for metformin in the context of chemo-radiation, with toxicity as the primary outcome.
  Patients in the Phase II trial will be assigned to a single arm (DL1), experimental treatment consisting of metformin plus chemo-radiation.
  Metformin: Metformin will be administered orally twice daily during treatment with chemo-radiation for head and neck squamous cell carcinoma. This will occur 7 to 11 days prior to chemotherapy and radiation.
  Dose Level 1 (DL1): 850 mg per os (PO) twice daily (BID)
- Single Arm, Treatment: DL2: Patients in the Phase I trial will be assigned to a single arm, experimental treatment which will test dose escalation for metformin in the context of chemo-radiation, with toxicity as the primary outcome.
  Patients in the Phase II trial will be assigned to a single arm (DL1), experimental treatment consisting of metformin plus chemo-radiation.
  Metformin: Metformin will be administered orally twice daily during treatment with chemo-radiation for head and neck squamous cell carcinoma. This will occur 7 to 11 days prior to chemotherapy and radiation.
  Dose Level 2 (DL2): 1500 mg per os (PO) twice daily (BID)
- Single Arm, Treatment: DL-1: Patients in the Phase I trial will be assigned to a single arm, experimental treatment which will test dose escalation for metformin in the context of chemo-radiation, with toxicity as the primary outcome.
  Patients in the Phase II trial will be assigned to a single arm (DL1), experimental treatment consisting of metformin plus chemo-radiation.
  Metformin: Metformin will be administered orally twice daily during treatment with chemo-radiation for head and neck squamous cell carcinoma. This will occur 7 to 11 days prior to chemotherapy and radiation.
  Dose Level -1 (DL-1): 500 mg per os (PO) twice daily (BID)
Period: Phase I
Arm/Group | Single Arm, Treatment: DL1 (Phase I) | Single Arm, Treatment: DL2 | Single Arm, Treatment: DL-1 | Single Arm, Treatment: DL1 (Phase II)
Started | 9 | 3 | 0 | 0
Completed | 7 | 2 | 0 | 0
Not Completed | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Period: Phase II
Arm/Group | Single Arm, Treatment: DL1 (Phase I) | Single Arm, Treatment: DL2 | Single Arm, Treatment: DL-1 | Single Arm, Treatment: DL1 (Phase II)
Started | 0 | 0 | 1 (All patients underwent a 2 week "lead-in" period in order to decrease the gastrointestinal toxicity associated with metformin. During this "lead-in" period, all patients started metformin at the dose of 500mg PO BID and increased to their assigned dose levels at the end of the "lead-in" period. One patient, however, did not complete the "lead-in" period and was taken off study due to protocol violation, hence the assignment of this patient to the "lead-in" dose, or DL-1.) | 12
Completed | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Single Arm, Treatment: DL1 (Phase I); Single Arm, Treatment: DL1 (Phase II): Patients in the Phase I trial will be assigned to a single arm, experimental treatment which will test dose escalation for metformin in the context of chemo-radiation, with toxicity as the primary outcome.
  Patients in the Phase II trial will be assigned to a single arm (DL1), experimental treatment consisting of metformin plus chemo-radiation.
  Metformin: Metformin will be administered orally twice daily during treatment with chemo-radiation for head and neck squamous cell carcinoma. This will occur 7 to 11 days prior to chemotherapy and radiation.
  Dose Level 1: 850 mg per os (PO) twice daily (BID)
- Single Arm, Treatment: DL2: Patients in the Phase I trial will be assigned to a single arm, experimental treatment which will test dose escalation for metformin in the context of chemo-radiation, with toxicity as the primary outcome.
  Patients in the Phase II trial will be assigned to a single arm (DL1), experimental treatment consisting of metformin plus chemo-radiation.
  Metformin: Metformin will be administered orally twice daily during treatment with chemo-radiation for head and neck squamous cell carcinoma. This will occur 7 to 11 days prior to chemotherapy and radiation.
  Dose Level 2: 1500 mg per os (PO) twice daily (BID)
- Single Arm, Treatment: DL-1: Patients in the Phase I trial will be assigned to a single arm, experimental treatment which will test dose escalation for metformin in the context of chemo-radiation, with toxicity as the primary outcome.
  Patients in the Phase II trial will be assigned to a single arm (DL1), experimental treatment consisting of metformin plus chemo-radiation.
  Metformin: Metformin will be administered orally twice daily during treatment with chemo-radiation for head and neck squamous cell carcinoma. This will occur 7 to 11 days prior to chemotherapy and radiation.
  Dose Level 1: 500 mg per os (PO) twice daily (BID)
- Total: Total of all reporting groups
Arm/Group | Single Arm, Treatment: DL1 (Phase I) | Single Arm, Treatment: DL2 | Single Arm, Treatment: DL-1 | Single Arm, Treatment: DL1 (Phase II) | Total
Number analyzed (Participants) | 9 | 3 | 1 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (7.5) | 69.0 (7.5) | 64.0 (0.0) | 58.6 (6.3) | 60.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1
  Male | 9 | 3 | 1 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 8 | 3 | 1 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 8 | 2 | 1 | 12 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Dose-Limiting Toxicity
Description: Dose limiting toxicities include diarrhea/gastrointestinal disturbance and hypoglycemia requiring dose reduction, and they will be measured for the time frame detailed above. Adverse Events (AE)s will be graded in accordance with the NCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE) http://ctep.cancer.gov/ reporting/ctc.html. If not described in the NCI-CTCAE, AEs will be graded according to their severity using the following criteria: grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (life threatening).
Time Frame: treatment duration plus 30 days following treatment (an average of 13 weeks)
Population: Participants were considered for Phase I toxicity (dose-limiting toxicity) evaluation if they were enrolled in the Phase I portion and took 70% or more of the study drug throughout the course of the trial. 9 out of 25 subjects (7 on DL1 (Phase I), 2 on DL2) met this criterion.
Measure: Number; unit: dose-limiting toxicities
Arm/Group | Single Arm, Treatment: DL1 (Phase I) | Single Arm, Treatment: DL2
Number analyzed (Participants) | 7 | 2
dose-limiting toxicities | 0 | 0

2. Primary Outcome: Phase II - Efficacy (Disease Response Rate)
Description: Response and progression will be evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST1.1) Committee [Eur J Cancer. 2009 Jan; 45(2):228-47]. Changes in only the largest diameter (uni-dimensional measurement) of the tumor lesions are used in the RECIST 1.1 criteria. For the purposes of this study, patients should be reevaluated for response following completion of treatment as per current institutional protocol for this disease site: 1) spiral contrast enhanced computed tomography (CECT) at 10 weeks following completion of treatment or 2) positron emission tomography (PET) at 12 weeks following completion of treatment. Per RECIST v1.1 criteria for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Disease response rate is defined as the percentage of patients with OR.
Time Frame: Treatment duration plus 8-12 weeks following treatment completion (up to 21 weeks total)
Population: Participants were considered for Phase II efficacy (disease response rate) evaluation if they were enrolled in the Phase II portion and took 70% or more of the study drug throughout the course of the trial. 7 out of 25 subjects (7 on DL1 (Phase II)) met this criterion.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Single Arm, Treatment: DL1 (Phase II)
Number analyzed (Participants) | 7
percentage of participants with response | 100.0 [59.0 to 100.0]

3. Secondary Outcome: Phase II - Progression Free Survival
Description: Measurement of time from date of study registration to date of documented radiographic recurrence/progression or death.
Time Frame: Date of study registration to recurrence/progression/death or up to 2 years following treatment completion, whichever comes first.
Population: Participants were considered for Phase II progression free survival evaluation if they were enrolled in the Phase II portion and took 70% or more of the study drug throughout the course of the trial. 7 out of 25 subjects (7 on DL1 (Phase II)) met this criterion.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Single Arm, Treatment: DL1 (Phase II)
Number analyzed (Participants) | 7
months | 22.7 [9.8 to 29.3]

4. Secondary Outcome: Phase II - Overall Survival
Description: Measurement of time from date of study registration to date of death.
Time Frame: Date of study registration to death or up to 2 years following treatment completion, whichever comes first.
Population: Participants were considered for Phase II overall survival evaluation if they were enrolled in the Phase II portion and took 70% or more of the study drug throughout the course of the trial. 7 out of 25 subjects (7 on DL1 (Phase II)) met this criterion.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Single Arm, Treatment: DL1 (Phase II)
Number analyzed (Participants) | 7
months | 22.7 [9.8 to 29.3]

ADVERSE EVENTS:
Time Frame: The AE collection/reporting period began with the first day of treatment with metformin and was completed at 30 days following treatment completion of each participant. This resulted in a 13 week period of AE collecting/reporting for each participant. All-cause mortality data was collected up to 2 years following treatment completion, as per Outcome Measure 4.
Groups:
- Single Arm, Treatment: DL-1: Patients in the Phase I trial will be assigned to a single arm, experimental treatment which will test dose escalation for metformin in the context of chemo-radiation, with toxicity as the primary outcome.
  Patients in the Phase II trial will be assigned to a single arm (DL1), experimental treatment consisting of metformin plus chemo-radiation.
  Metformin: Metformin will be administered orally twice daily during treatment with chemo-radiation for head and neck squamous cell carcinoma. This will occur 7 to 11 days prior to chemotherapy and radiation.
  Dose Level -1: 500 mg per os (PO) twice daily (BID)
Arm/Group | Single Arm, Treatment: DL1 (Phase I) | Single Arm, Treatment: DL2 | Single Arm, Treatment: DL-1 | Single Arm, Treatment: DL1 (Phase II)
All-Cause Mortality (participants affected / at risk) | 4/9 | 2/3 | 0/1 | 4/12
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/3 | 0/1 | 3/12
Other Adverse Events (participants affected / at risk) | 8/9 | 3/3 | 1/1 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm, Treatment: DL1 (Phase I) (N=9) | Single Arm, Treatment: DL2 (N=3) | Single Arm, Treatment: DL-1 (N=1) | Single Arm, Treatment: DL1 (Phase II) (N=12)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | NA | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | NA | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | NA | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | NA | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | NA | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | NA | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | NA | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | NA | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | NA | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm, Treatment: DL1 (Phase I) (N=9) | Single Arm, Treatment: DL2 (N=3) | Single Arm, Treatment: DL-1 (N=1) | Single Arm, Treatment: DL1 (Phase II) (N=12)
Anemia (Blood and lymphatic system disorders) | 7 (13) | 3 (5) | 1 (2) | 7 (18)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 3 (5) | 0 (0) | 5 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (8)
Dysphagia (Gastrointestinal disorders) | 6 (7) | 1 (1) | 0 (0) | 6 (13)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (6) | 1 (1) | 1 (1) | 9 (11)
Nausea (Gastrointestinal disorders) | 7 (11) | 3 (3) | 1 (1) | 6 (9)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7) | 1 (1) | 0 (0) | 2 (3)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (4)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 5 (6)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 2 (2) | 1 (2) | 0 (0) | 5 (9)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Lymphocyte count decreased (Investigations) | 4 (11) | 2 (2) | 0 (0) | 5 (14)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 3 (5)
Platelet count decreased (Investigations) | 2 (2) | 2 (3) | 0 (0) | 5 (12)
Weight loss (Investigations) | 4 (6) | 2 (3) | 1 (1) | 8 (18)
White blood cell decreased (Investigations) | 2 (4) | 2 (3) | 1 (1) | 6 (12)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0) | 6 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 2 (5) | 1 (2) | 7 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (7)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 1 (1) | 10 (18)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (10)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 9 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT02949700/Prot_SAP_000.pdf